CLINICAL TRIAL: NCT00528281
Title: A Single-arm, Two-stage Phase II Study of Lapatinib and Pemetrexed in the Second Line Treatment of Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Phase II Trial of Lapatinib (TYKERB) + Pemetrexed (ALIMTA) in Advanced Non Small Cell Lung Cancer With an Initial Dose Finding Phase
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF109462
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Non Small Cell Lung Cancer (NSCLC); Pemetrexed,; Lapatinib (GW572016),
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Lapatinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lapatinib + pemetrexed (Experimental): This is a single-arm, two-stage, multicenter Phase II study to determine the clinical activity of pemetrexed with lapatinib.
  Interventions: Drug: Lapatinib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Lapatinib — Lapatinib was administered once daily orally. Patients will begin treatment at Dose Level 0, using a lower dose of pemetrexed, 400mg (approved dose is 500mg). Absent a DLT or need for treatment delay in cycle 1, Dose level 0 or 1, patients may be dose escalated to dose level 1 or 2, respectively in cycle 2.
Drug: Pemetrexed — Pemetrexed is administered intravenously on a 21 day schedule. Two dose levels are used in the dose escalation: 400 and 500 mg.

SUMMARY:
This phase II study is a single-arm, two-stage, multicentre study to determine the clinical activity of lapatinib in combination with pemetrexed in patients with Non-Small Cell Lung Cancer (NSCLC) who have received one prior cytotoxic chemotherapy regimen. There will be a short safety run in portion of the study to determine the optimal treatment regimen (OTR) for the combination, since these two drugs have not previously been used together.

Approximately 27 patients will be enrolled into the first stage of the study and if sufficient responses are seen an additional 27 patients will be enrolled into the second stage giving an overall evaluable patient number of 54. Patients will be treated with pemetrexed plus lapatinib at the determined OTR to disease progression, death or withdrawal from the study treatment for any reason.

Safety and efficacy assessments will be performed on all patients at 6-week intervals, as well as at the end of treatment. Patients withdrawn from study treatment with stable disease will be assessed every 6 weeks until progression. Thereafter, patients will be followed for survival at approximately 12-week intervals until death or to a maximum of 5 years after last patient is enrolled, whichever comes first.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed informed consent;
* Patients must be 18 years old;
* Subjects must have stage IIIB or IV NSCLC .
* Recurrent or persistent NSCLC following one previous line of cytotoxic chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2;
* Life expectancy of 12 weeks;
* Have adequate organ function baseline laboratory values for inclusion;

EXCLUSION CRITERIA:

* History of other malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible;
* Known history of or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or antiseizure medication for = 3 months prior to study enrollment.
* Peripheral neuropathy of grade 3 or higher;
* Concurrent cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, and tumor embolization).
* Prior exposure to pemetrexed or an EGFR inhibitor in combination with 5-FU or a 5FU prodrug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09-20 (Actual); Primary Completion 2009-05-27 (Actual); Study Completion 2009-05-27 (Actual)

PRIMARY OUTCOMES:
OTR of the combination of lapatinib and pemetrexed

SECONDARY OUTCOMES:
anti-tumour activity of lapatinib in terms of overall response rate
anti-tumour activity of lapatinib in terms of duration of response, time to response, time to progression, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (2):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- GSK Investigational Site, Orbassano (TO), Piedmont, Italy
- GSK Investigational Site, Poznan, Poland
- GSK Investigational Site, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Background] Ramlau R, Thomas M, Novello S, Plummer R, Reck M, Kaneko T, Lau MR, Margetts J, Lunec J, Nutt J, Scagliotti GV. Phase I Study of Lapatinib and Pemetrexed in the Second-Line Treatment of Advanced or Metastatic Non-Small-Cell Lung Cancer With Assessment of Circulating Cell Free Thymidylate Synthase RNA as a Potential Biomarker. Clin Lung Cancer. 2015 Sep;16(5):348-57. doi: 10.1016/j.cllc.2015.01.004. Epub 2015 Jan 20. PMID 25700774
- See also: Results for study EGF109462 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/EGF109462?search=study&search_terms=109462#rs